CLINICAL TRIAL: NCT00298220
Title: Engaging General Practice in the Prevention of Patients With Alcohol Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: KWAZO/GPA-01; 50-50115-98-041
Record Dates: First submitted 2006-02-21; First posted 2006-03-01 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-08

CONDITIONS: Alcohol Drinking
Keywords: Family Practice; Intervention Studies; Prevention and Control
MeSH Terms: conditions — Alcohol Drinking

ARMS (2):
- training (Active Comparator): tailored multi-component implementation program
  Interventions: Behavioral: Feedback about patients at risk; Behavioral: Dissemination guideline and patient information letters; Behavioral: Tailored educational training; Behavioral: Tailored outreach based facilitator support; Behavioral: Facilitation of co-operation with local addiction services; Behavioral: Patient directed interventions; Behavioral: Reminder-card for GP's desk; Behavioral: Personal feedback to patients
- control (No Intervention)
  Interventions: Behavioral: Feedback about patients at risk; Behavioral: Dissemination guideline and patient information letters; Behavioral: Personal feedback to patients

INTERVENTIONS:
Behavioral: Feedback about patients at risk — GPTs receive this feedback about their patient population; obtained through premeasurement results
Behavioral: Dissemination guideline and patient information letters
Behavioral: Tailored educational training — for GP(T)s
  Arms: training
Behavioral: Tailored outreach based facilitator support — in the practices of the GPTs
  Arms: training
Behavioral: Facilitation of co-operation with local addiction services
  Arms: training
Behavioral: Patient directed interventions — Like poster for the waiting room, self-help booklets, folders
  Arms: training
Behavioral: Reminder-card for GP's desk
  Arms: training
Behavioral: Personal feedback to patients — Patients receive advise based on their premeasurement answers

SUMMARY:
The aim of the study is to test whether or not a tailored multi-component intervention program to increase the activity of general practice teams in the prevention of hazardous and harmful alcohol consumption results in increase advice giving rate to patient with hazardous and harmful alcohol consumption and a better patient outcome in terms of hazardous and harmful alcohol consumption.

The primary objectives of the proposed study are:

1. to test the (cost) effectiveness of a tailored multi-component implementation program to engage general practices (i.e. GPs, nurse practitioners or practice nurses/assistants) in the prevention of hazardous or harmful alcohol consumption, changing both providers' advice giving behaviour and patients' alcohol consumption
2. to identify predictors of effect
3. to examine whether or not the implementation of a tailored multi-component implementation program to engage general practice in the prevention of hazardous or harmful alcohol consumption is feasible.

DETAILED DESCRIPTION:
Hazardous and harmful alcohol consumption is likely to cause damage to health, either physical or mental. The prevention of harmful alcohol consumption results in a reduction of alcohol related diseases, of emergency and hospital use, and of societal related problems, and it results in direct health care savings as well as in non-health care savings. General practice is an important setting to intervene with patients whose drinking is hazardous or harmful to their health. Despite the evidence for the efficacy and cost effectiveness of case finding and brief interventions in general practice, such interventions are rarely integrated into routine practice. Based on the literature it is recommended to develop a tailored multi-component implementation program to engage general practice in the prevention of patients with alcohol consumption.

In our trial such a tailored multi-component intervention program is offered to the general practice team (GPT). The participants in our trial are the GPT, not the patients. The GPTs practising in Mid-West and Mid-South are invited to participate in the trial by an invitational letter, including an information leaflet. Participation is not obligatory, but based on own interest of the GPT. Next, GPTs who are willing to participate in the trial are random allocated to the intervention or control condition. Besides the effect outcome measures described in the 'Outcome measure" part there are process and costs measures described.

Besides measurements at the GPT-level, we also conduct measurements at the patient level. All patients of 18 years or older visiting the GPT during a pre-defined 3-month period are asked to fill in the Alcohol Use Disorders identification Test (AUDIT). This measurement takes place before the intervention starts. Only those patients at risk are asked to fill in the AUDIT after the intervention ended. As described in the 'Outcome part', the AUDIT is used to describe the effects of the intervention program at the patient level. Patients receive individual feedback with personal advice depending on their AUDIT score. Patients are not informed about whether the GPT is allocated to the intervention program or control condition (usual care) (single blind).

Comparison: GPTs participated in the multi-component intervention program (see Interventions; intervention group) are compared to GPTs who didn't participate in the multi-component intervention program (control group). The GPTs in the control group receive the NHG guideline and NHG patient information letters, which can be seen as usual care. In addition the receive feedback about the number of patients at risk because of their alcohol consumption, which can be seen as a minimal intervention.

ELIGIBILITY:
Inclusion Criteria:

* GP
* all GPs in a GPT have to participate or
* patients should be listed per GP

There are no exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-07; Primary Completion 2008-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
- Proportion of patients who, with an initial AUDIT score of 16 or more, have an AUDIT score at follow-up (= 18 months) of 15 or less.
- Proportion of patients who, with an initial AUDIT score of 16 or more, have been given advice by the general practitioner or by other staff (e.g. nurse practitioner, practice nurse).

SECONDARY OUTCOMES:
- Average AUDIT score at follow-up (= 18 months).
- Average alcohol consumption as measured by the AUDIT at follow-up (= 18 months).
- Proportion of patients with hazardous or harmful alcohol consumption as measured by the AUDIT at follow-up (= 18 months).
- Proportion of patients with harms from alcohol as measured by the AUDIT at follow-up (= 18 months).
- Proportion of patients with alcohol dependence as measured by the AUDIT at follow-up (= 18 months).
- Average SAAPPQ score.
- Change in SAAPPQ score.

CONTACTS AND LOCATIONS:
Overall Officials: M. Laurant, PhD, Principal Investigator — Centre for Quality for Care Research Nijmegen

REFERENCES:
- [Background] Lemmens PH. Relationship of alcohol consumption and alcohol problems at the population level. In Heather N, Peters TJ, Stockwell T (eds). International handbook of alcohol dependence and problems. Chischester: John Wiley & Sons, Ltd. 2001
- [Background] Anderson P, Cremona A, Paton A, Turner C, Wallace P. The risk of alcohol. Addiction. 1993 Nov;88(11):1493-508. doi: 10.1111/j.1360-0443.1993.tb03135.x. PMID 8286995
- [Background] Anderson P. Alcohol and risk of physical harm. In Holder HD & Edwards G (eds). Alcohol and public policy: evidence and issues. Oxford: Oxford Medical Publications. 1995
- [Background] Guilbert JJ. The world health report 2002 - reducing risks, promoting healthy life. Educ Health (Abingdon). 2003 Jul;16(2):230. doi: 10.1080/1357628031000116808. No abstract available. PMID 14741909
- [Background] Garretsen HFL, Knibbe RA. Alcohol prevalentie onderzoek Rotterdam/Limburg. Landelijk eindrapport. Rijswijk: Ministerie van WVC. 1983
- [Background] Volksgezondheid Toekomst Verkenning. Natioaal Kompas Volksgezondheid. Bilthoven: RIVM, http://www.nationaal kompas.nl, versie 2.4, september 2003
- [Background] Cornel M et al. NHG Standaard M10. Problematisch alcoholgebruik. Huisarts en Wetenschap 1998; 41 (12): 582-90
- [Background] Ministerie van VWS. Zorgnota 2003
- [Background] Anderson P. The effectiveness of general practitioners' advice in reducing the risk of alcohol. IN: Neil A et al (eds). Prevention of Cardiovascular Disease: An evidence-based approach. 2nd Ed. Oxford: Oxford University Press. In press
- [Background] Sutherland G. Smoking cessation: Evidence for counseling efficacy. J of Clinical Psychiatry. In press
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Benefit-cost analysis of brief physician advice with problem drinkers in primary care settings. Med Care. 2000 Jan;38(1):7-18. doi: 10.1097/00005650-200001000-00003. PMID 10630716
- [Background] Spandorfer JM, Israel Y, Turner BJ. Primary care physicians' views on screening and management of alcohol abuse: inconsistencies with national guidelines. J Fam Pract. 1999 Nov;48(11):899-902. PMID 10907628
- [Background] Anderson P, Laurant M, Kaner E, Wensing M, Grol R. Engaging general practitioners in the management of hazardous and harmful alcohol consumption: results of a meta-analysis. J Stud Alcohol. 2004 Mar;65(2):191-9. doi: 10.15288/jsa.2004.65.191. PMID 15151349
- [Background] Murphy HB. Hidden barriers to the diagnosis and treatment of alcoholism and other alcohol misuse. J Stud Alcohol. 1980 May;41(5):417-28. doi: 10.15288/jsa.1980.41.417. PMID 7412295
- [Background] Skinner HA, Holt S. Early intervention for alcohol problems. J R Coll Gen Pract. 1983 Dec;33(257):787-91. PMID 6361249
- [Background] Hulscher ME, Wensing M, Grol RP, van der Weijden T, van Weel C. Interventions to improve the delivery of preventive services in primary care. Am J Public Health. 1999 May;89(5):737-46. doi: 10.2105/ajph.89.5.737. PMID 10224987
- [Background] Bero LA, Grilli R, Grimshaw JM, Harvey E, Oxman AD, Thomson MA. Closing the gap between research and practice: an overview of systematic reviews of interventions to promote the implementation of research findings. The Cochrane Effective Practice and Organization of Care Review Group. BMJ. 1998 Aug 15;317(7156):465-8. doi: 10.1136/bmj.317.7156.465. No abstract available. PMID 9703533
- [Background] Eccles M, Grimshaw J, Campbell M, Ramsay C. Research designs for studies evaluating the effectiveness of change and improvement strategies. Qual Saf Health Care. 2003 Feb;12(1):47-52. doi: 10.1136/qhc.12.1.47. PMID 12571345
- [Background] Moyer A, Finney JW, Swearingen CE, Vergun P. Brief interventions for alcohol problems: a meta-analytic review of controlled investigations in treatment-seeking and non-treatment-seeking populations. Addiction. 2002 Mar;97(3):279-92. doi: 10.1046/j.1360-0443.2002.00018.x. PMID 11964101
- [Background] Babor TF, et al. The Alcohol Use Disorders Identification Test Guidelines for Use in Primary Care. Geneva: World Health Organization WHO/MSD/MSB/01.6a.
- [Background] Anderson P, Kaner E, Wutzke S, Wensing M, Grol R, Heather N, Saunders J; World Health Organization Brief Intervention Study Group. Attitudes and management of alcohol problems in general practice: descriptive analysis based on findings of a World Health Organization international collaborative survey. Alcohol Alcohol. 2003 Nov-Dec;38(6):597-601. doi: 10.1093/alcalc/agg119. PMID 14633648
- [Background] Anderson P, Clement S. The AAPPQ revisited: the measurement of general practitioners' attitudes to alcohol problems. Br J Addict. 1987 Jul;82(7):753-9. doi: 10.1111/j.1360-0443.1987.tb01542.x. No abstract available. PMID 3478065
- [Background] Fiellin DA, Reid MC, O'Connor PG. Screening for alcohol problems in primary care: a systematic review. Arch Intern Med. 2000 Jul 10;160(13):1977-89. doi: 10.1001/archinte.160.13.1977. PMID 10888972
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Babor TF, Grant M, Acuda W, Burns FH, Campillo C, Del Boca FK, Hodgson R, Ivanets NN, Lukomskya M, Machona M, et al. A randomized clinical trial of brief interventions in primary care: summary of a WHO project. Addiction. 1994 Jun;89(6):657-60; discussion 660-78. doi: 10.1111/j.1360-0443.1994.tb00944.x. No abstract available. PMID 8069168
- [Background] Kaner E, Lock C, Heather N, McNamee P, Bond S. Promoting brief alcohol intervention by nurses in primary care: a cluster randomised controlled trial. Patient Educ Couns. 2003 Nov;51(3):277-84. doi: 10.1016/s0738-3991(02)00242-2. PMID 14630384
- [Background] Gross PA, Greenfield S, Cretin S, Ferguson J, Grimshaw J, Grol R, Klazinga N, Lorenz W, Meyer GS, Riccobono C, Schoenbaum SC, Schyve P, Shaw C. Optimal methods for guideline implementation: conclusions from Leeds Castle meeting. Med Care. 2001 Aug;39(8 Suppl 2):II85-92. PMID 11583124
- [Background] Grol R, Jones R. Twenty years of implementation research. Fam Pract. 2000 Feb;17 Suppl 1:S32-5. doi: 10.1093/fampra/17.suppl_1.s32. No abstract available. PMID 10735266
- [Background] Grol R. Successes and failures in the implementation of evidence-based guidelines for clinical practice. Med Care. 2001 Aug;39(8 Suppl 2):II46-54. doi: 10.1097/00005650-200108002-00003. PMID 11583121
- [Background] van Bokhoven MA, Kok G, van der Weijden T. Designing a quality improvement intervention: a systematic approach. Qual Saf Health Care. 2003 Jun;12(3):215-20. doi: 10.1136/qhc.12.3.215. PMID 12792013
- [Background] Prochaska JO, Di Clemente CC. The transtheoretical approach: crossing traditional boundaries of therapy. Homewood, IL: Dow Jones-Irwin. 1984
- [Background] Rogers EM. Diffusion of innovations. 4th ed. New York: Free Press. 1995
- [Background] Fishbein M, Ajzen I. Belief, attitude, intentention and behavior: an introduction to therory and research. Reading, MA: Addison Wesley, 1975
- [Background] Mc Guire WJ. Attitudes an attitude change. In: Lindzey G, Aronson E (eds). The handbook of social psychology. New York: Random House, 1985; 233-346
- [Background] Anderson P, Jane-Llopis E. How can we increase the involvement of primary health care in the treatment of tobacco dependence? A meta-analysis. Addiction. 2004 Mar;99(3):299-312. doi: 10.1111/j.1360-0443.2003.00672.x. PMID 14982543
- [Background] Davis D, O'Brien MA, Freemantle N, Wolf FM, Mazmanian P, Taylor-Vaisey A. Impact of formal continuing medical education: do conferences, workshops, rounds, and other traditional continuing education activities change physician behavior or health care outcomes? JAMA. 1999 Sep 1;282(9):867-74. doi: 10.1001/jama.282.9.867. PMID 10478694
- [Background] Hulscher ME, van Drenth BB, van der Wouden JC, Mokkink HG, van Weel C, Grol RP. Changing preventive practice: a controlled trial on the effects of outreach visits to organise prevention of cardiovascular disease. Qual Health Care. 1997 Mar;6(1):19-24. doi: 10.1136/qshc.6.1.19. PMID 10166597
- [Background] Lobo CM, Frijling BD, Hulscher ME, Bernsen RM, Braspenning JC, Grol RP, Prins A, van der Wouden JC. Improving quality of organizing cardiovascular preventive care in general practice by outreach visitors: a randomized controlled trial. Prev Med. 2002 Nov;35(5):422-9. doi: 10.1006/pmed.2002.1095. PMID 12431890
- [Background] Fullard E, Fowler G, Gray M. Promoting prevention in primary care: controlled trial of low technology, low cost approach. Br Med J (Clin Res Ed). 1987 Apr 25;294(6579):1080-2. doi: 10.1136/bmj.294.6579.1080. PMID 3107700
- [Background] Astrop P. Facilitator--the birth of a new profession. Health Visit. 1988 Oct;61(10):311-2. No abstract available. PMID 3198412
- [Background] Hulscher MEJL. Implementing prevention in general practice: a study on cardiovascular disease. Doctoral thesis. Nijmegen: 1998
- [Background] Huiberts A, Boon B. Alcoholadvies op maat online. G: vakblad over gezondheid en maatschappij 2003; 1: 28-9
- [Background] Riper H, Kramer, J Effectiviteit van een zelfhulpboekje voor probleemdrinkers. Utrecht: Trimbos-instituut. In preparation
- [Background] Hermens R. Cervical cancer screening. Quality improvement interventions in general practice. Doctoral thesis. Nijmegen: 2003
- [Background] Whitfield JB. Diagnostic and monitoring investigations. In: Heather N, et al (eds.) International handbook of alcohol dependence and problems. Chichester: John Wiley & Sons, Ltd., (2001).
- [Derived] Keurhorst M, van Beurden I, Anderson P, Heinen M, Akkermans R, Wensing M, Laurant M. GPs' role security and therapeutic commitment in managing alcohol problems: a randomised controlled trial of a tailored improvement programme. BMC Fam Pract. 2014 Apr 17;15:70. doi: 10.1186/1471-2296-15-70. PMID 24742032
- [Derived] van Beurden I, Anderson P, Akkermans RP, Grol RP, Wensing M, Laurant MG. Involvement of general practitioners in managing alcohol problems: a randomized controlled trial of a tailored improvement programme. Addiction. 2012 Sep;107(9):1601-11. doi: 10.1111/j.1360-0443.2012.03868.x. Epub 2012 May 8. PMID 22372573